CLINICAL TRIAL: NCT00937183
Title: Vaccination of Lymphoma Patients With Dendritic Cell-lymphoma Cell Hybrids and Dendritic Cells Pulsed With Tumor Lysates
Brief Title: Dendritic Cell Vaccine in Treating Patients With Indolent B-Cell Lymphoma or Multiple Myeloma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jan Walewski (Other)
Responsible Party: Sponsor-Investigator, Jan Walewski, Head, Dept. of Lymphoid Malignancies, Maria Sklodowska-Curie National Research Institute of Oncology
Organization: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSCMI-40-2003; CDR0000636859 (Registry Identifier: PDQ (Physician Data Query)); EU-20913
Record Dates: First submitted 2009-07-08; First posted 2009-07-10 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm
Keywords: dendritic cell vaccine; tumor cell lysate; lymphoma
MeSH Terms: conditions — Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell

INTERVENTIONS:
Biological: autologous lymphoma cell lysate-pulsed autologous dendritic cell vaccine
Biological: autologous lymphoma cell/allogeneic dendritic cell electrofusion hybrid vaccine
Biological: autologous lymphoma cell/autologous dendritic cell electrofusion hybrid vaccine

SUMMARY:
RATIONALE: Biological therapies, such as a dendritic cell vaccine made with a patient's cancer cells, may stimulate the immune system in different ways and stop cancer cells from growing.

PURPOSE: This phase I/II trial is studying the side effects of dendritic cell vaccine and to see how well it works in treating patients with indolent B-cell lymphoma or multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluation of feasibility of dendritic cell (DC)-based vaccination program using autologous tumor cells and/or lysates in patients with indolent B cell lymphomas or multiple myeloma as an adjuvant therapy to induce immune response in remission after cytoreductive treatment.
* Evaluation of the immune response of patients treated with this regimen.
* Evaluation the progression-free survival of patients treated this regimen.
* Evaluate the adverse events of this regimen in these patients.

OUTLINE: Patients receive intranodal (under ultrasound guidance) or subcutaneous vaccinations of adjuvant electrofusion hybrids of autologous dendritic cells (DC) with autologous lymphoma cells, electrofusion hybrids of allogeneic DC with autologous lymphoma cells, and/or autologous DC pulsed with autologous tumor lysate cells in weeks 0, 2, 4, 8, 12, 18, 26, and 50.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of 1 of the following:

  * Mantle cell lymphoma
  * Marginal zone lymphoma
  * Follicular lymphoma
  * Small lymphocytic lymphoma/chronic lymphocytic leukemia
  * Multiple myeloma
  * Lymphoplasmacytic lymphoma/Waldenström macroglobulinemia
  * Diffuse large B-cell lymphoma
* Adequate sample size and lymphoma cell content in the fresh tissue collected
* No bulky or progressive disease

PATIENT CHARACTERISTICS:

* Life expectancy > 3 months
* No evidence of lung, heart, liver, or renal failure or severe neurologic disorder
* No autoimmune disease or atopic allergy
* No HIV positivity
* No other malignancy

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2003-09; Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Immune response
Progression-free survival
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jan Walewski, MD, Study Chair — Maria Sklodowska-Curie National Research Institute of Oncology
Locations (1):
- Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology - Warsaw, Warsaw, Poland